CLINICAL TRIAL: NCT05085730
Title: Clinical Assessment of Skin Quality and Efficacy of Dermal Line Improvement Following Four Bipolar Radiofrequency Microneedling Treatments
Brief Title: Assessment Skin Quality and Efficacy of Dermal Line After Four Bipolar Radiofrequency Microneedling Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey M. Kenkel, Principle Investigator, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 2021-0916
Record Dates: First submitted 2021-09-27; First posted 2021-10-20 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Aging
Keywords: skin aging; bipolar radiofrequency; microneedling; dermal lines

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental): All subjects will receive 4 separate treatments with the InMode Morpheus8 System.
  Interventions: Device: InMode Morpheus8 System

INTERVENTIONS:
Device: InMode Morpheus8 System — The InMode Morpheus8 System is a bipolar fractional radiofrequency device which uses microneedles and thermal heat to stimulate neocollagenesis and neoelastogenesis.

SUMMARY:
This study intends to evaluate the safety and effectiveness of the InMode Morpheus8 System to treat facial and neck skin and assess its effect on skin quality and dermal lines. This device has been FDA cleared for full body subdermal adipose tissue remodeling.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and efficacy of a bipolar fractional radiofrequency treatment via use of the InMode Morpheus8 System to achieve skin texture and quality change and to treat facial fine lines and wrinkles of the lower face.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female adults between ages 21-70 years of age.
2. Presence of facial dermal lines and skin changes of the lower face associated with age or environmental exposure.
3. Confirmed BMI ≤ 35.
4. Subjects who can read, understand, and sign the Informed Consent Form.
5. Subjects willing and able to comply with all study requirements.
6. Fitzpatrick skin type I-VI.
7. Minimum of 1 on the Lemperle Wrinkle Assessment Scale, Allergan Fine Line Scale and Allergan Skin Roughness Scale
8. Subject is willing not to undergo any type of aesthetic procedure that could confound the study device treatment effects until he/she completes the study.

Exclusion Criteria:

1. Active localized or systemic infections, that may alter wound healing.
2. Immunocompromised subjects.
3. Subjects with coagulation disorder.
4. History of skin photosensitivity disorders, or use of photosensitizing drugs (e.g., tetracycline or sulfa drugs).
5. Pregnant and/or lactating (All female volunteers will be advised about using birth control during the period of study).
6. 5 on the Lemperle Wrinkle Assessment Scale or 4 on the Allergan Fine Line Scale and/or Allergan Skin Roughness Scales
7. Scarring in areas to be treated.
8. Tattoos in the treatment areas to be treated.
9. Significant open facial wounds or lesions.
10. Severe or cystic acne in treatment areas.
11. Current active smoker.
12. Use of Accutane (Isotretinoin) within the past 6 months.
13. Use of topical retinoids within 48 hours.
14. Use of prescription anticoagulants.
15. Pacemaker or internal defibrillator.
16. History of skin disorders resulting in abnormal wound healing (i.e. keloids, extreme dry and fragile skin).
17. Subjects on current oral corticosteroid therapy or within the past 6 months
18. Metal implants in the treatment area.
19. In the opinion of the investigator, subject is unwilling or unable to adhere to all study requirements, including application and follow-up visits.
20. Subjects with a history of radiation therapy to the treatment area.
21. Subject has a history of allergy to lidocaine or ester-based local anesthetics.
22. Subjects with significant cardiac history or rhythm disturbance who may be unable to tolerate lidocaine with epinephrine.
23. Subjects with any skin pathology or condition in the treatment area that could interfere with evaluation or with the use of typical ancillary medical treatments or care used before, during or after treatments (e.g. psoriasis, rosacea, eczema, seborrheic dermatitis, vitiligo, hyper or hypo-skin pigmentation conditions such as post inflammatory hyperpigmentation).
24. Subjects who are unwilling to shave excessive hair in the treatment area that might influence or impair evaluation in the opinion of the Investigator.
25. Subjects have undergone skin resurfacing or tightening treatments in the treatment area over the past year.
26. Subjects have undergone dermatological treatments such as fillers and neurotoxins for the past 6 months in the treatment area.
27. Subjects have undergone laser and light treatments in the treatment area over the past 3 months.
28. Subjects have undergone superficial peel or microdermabrasion within 4 weeks.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Kenkel, MD, Principal Investigator — UT Southwestern- Department of Plastic Surgery
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 13
Completed | 8
Not Completed | 5
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change of Fine Lines and Wrinkles
Description: Lemperle Wrinkle Assessment Scale- wrinkling will be assessed according to scales definitions.
  0- No wrinkles
  1. Just perceptible wrinkles
  2. Shallow wrinkles
  3. Moderately thick wrinkles
  4. Deep wrinkles, well defined edges
  5. Very deep wrinkles, redundant folds
  Lower value would indicate improvement.
Time Frame: Baseline, 3 Months and 6 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline; Month 3; Month 6: All subjects will receive 4 separate treatments with the InMode Morpheus8 System.
  InMode Morpheus8 System: The InMode Morpheus8 System is a bipolar fractional radiofrequency device which uses microneedles and thermal heat to stimulate neocollagenesis and neoelastogenesis.
Arm/Group | Baseline | Month 3 | Month 6
Number analyzed (Participants) | 8 | 8 | 8
score on a scale
  Nasolabial Fold | 1.25 (0.71) | 1.625 (1.06) | 1 (0.93)
  Upper Lip Lines | 1.56 (0.50) | 1.75 (0.89) | 1.125 (0.64)
  Corner of Mouth Lines | 2.13 (1.36) | 1.5 (1.20) | 1.25 (1.04)
  Marionette Lines | 1.25 (1.39) | 1.31 (1.03) | 1.06 (1.08)
  Lower Lip Line | 1.06 (0.56) | 1.25 (0.89) | 0.5 (0.53)

2. Primary Outcome: Change of Fine Lines
Description: Allergan Scale for Fine Lines- fine lines of the midface/cheeks will be assessed according to the scales definition.
  0- None
  1. Minimal (1-2 superficial lines)
  2. Moderate (3-5 superficial lines)
  3. Severe (<5 superficial lines; no crosshatching)
  4. Diffuse (diffuse superficial lines; crosshatching)
  Lower value would indicate improvement
Time Frame: Baseline, 3 Months and 6 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | Month 3 | Month 6
Number analyzed (Participants) | 8 | 8 | 8
score on a scale | 1.625 (0.518) | 2 (0.532) | 1.375 (0.916)

3. Primary Outcome: Change of Skin Roughness
Description: Allergan Skin Roughness Scale Assessment- roughness will be assessed according to the scaled definitions based on skin coarseness, crosshatching and elastosis in midface area.
  0- None (smooth visual skin texture)
  1. Minimal (slightly course and uneven visual skin texture)
  2. Moderate (Moderately coarse and uneven visual skin texture; early elastosis)
  3. Severe (severe coarse visual skin texture, crosshatching lines; some elastosis)
  4. Diffuse (extreme coarse visual skin texture, deep crosshatched creases; extreme elastosis)
  Lower value would indicate improvement
Time Frame: Baseline, 3 Months and 6 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | Month 3 | Month 6
Number analyzed (Participants) | 8 | 8 | 8
score on a scale | 1.25 (0.71) | 0.5 (0.76) | 0.38 (0.75)

4. Primary Outcome: Global Aesthetic Improvement Scale (GAIS)
Description: Scale will be used to assess aesthetic change
  1. Very much improved
  2. Much improved
  3. Improved
  4. No Change
  5. Worse
  Lower value would indicate improvement
Time Frame: 3 Months and 6 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Month 3 | Month 6
Number analyzed (Participants) | 8 | 8
units on a scale
  Clinician GAIS (Live Assessment) | 3.81 (0.84) | 2.38 (1.06)
  Subject GAIS (Live Assessment) | 2.88 (0.99) | 2.63 (1.06)
  Clinician GAS (Photo Assessment) | 3.81 (0.55) | 3.25 (0.57)

5. Secondary Outcome: Adverse Events
Description: Adverse events will be monitored at each visit
Time Frame: Baseline, Day 30, Day 60, Day 90, Month 3 and Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 13
Participants | 0

6. Secondary Outcome: Change in Exploratory Thickness/Density- High Resolution Ultrasound
Description: high resolution ultrasound will be utilized to assess skin thickness/density.
Time Frame: Baseline, 3 Months and 6 Months
Population: 13 pts originally enrolled in the study- 5 subjects withdrew consent.
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Baseline | Month 3 | Month 6
Number analyzed (Participants) | 8 | 8 | 8
μm
  Epidermal Thickness | 72 (7.07) | 82.67 (15.02) | 73 (8.90)
  Epidermal Density | 69.53 (11.02) | 73.30 (38.51) | 79.65 (19.43)
  Dermal Thickness | 1257.33 (351.80) | 1214.83 (186.151) | 1311.33 (175.08)
  Dermal Density | 10.94 (4.88) | 17.18 (11.54) | 21.32 (9.66)

7. Secondary Outcome: Change in Barrier Skin Function- TEWL
Description: Transepidermal Water Loss Measurements (TEWL measurements) (via Bio Aquaflux) will be used to evaluate barrier function of the skin epidermal layer after treatments. It is used to assess skin thickness, density, firmness as well as the integrity of the stratum corneum. Skin barrier dysfunction results in increased TEWL.
Time Frame: Baseline, 3 Months and 6 Months
Population: Overall 13 pts enrolled in the study and 5 withdrew consent. An additional subject did not have a measurement obtained during their final visit thus was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: g/m^2/h
Arm/Group | Baseline | Month 3 | Month 6
Number analyzed (Participants) | 7 | 7 | 7
g/m^2/h | 26.16 (4.97) | 22.51 (6.87) | 18.08 (2.81)

8. Secondary Outcome: Biomechanical Tissue Measurements (Laxity, Elasticity)
Description: Bio-Mechanical Tissue Characterization (BTC2000) is a laser measurement system for objective, quantitative and sensitive analyses of the bio-mechanical properties of: Skin to assess skin thickness, density, firmness as well as the integrity of the stratum corneum.
Time Frame: Baseline, 3 Months and 6 Months
Population: Overall 13 pts consented for this study but 5 withdrew consent.
Measure: Mean (Standard Deviation); unit: mm/%
Arm/Group | Baseline | Month 3 | Month 6
Number analyzed (Participants) | 8 | 8 | 8
mm/%
  Laxity | 1.05 (0.40) | 0.66 (0.33) | 0.89 (0.29)
  Elasticity | 0.69 (0.24) | 0.54 (0.22) | 0.54 (0.23)

9. Secondary Outcome: Biomechanical Tissue Measurements (Elastic, Viscoelastic and Ultimate Deformation)
Description: as for outcome 8
Time Frame: Baseline, 3 Months and 6 Months
Population: Overall 13 pts consented for this study but 5 withdrew consent.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Baseline | Month 3 | Month 6
Number analyzed (Participants) | 8 | 8 | 8
mm
  Elastic Deformation | 1.57 (0.43) | 1.1 (0.36) | 1.23 (0.31)
  Viscoelastic Deformation | 0.10 (0.03) | 0.07 (0.02) | 0.07 (0.02)
  Ultimate Deformation | 1.66 (0.45) | 1.17 (0.36) | 1.34 (0.32)

10. Secondary Outcome: Biomechanical Tissue Measurements (Stiffness)
Description: as for outcome 8
Time Frame: Baseline, 3 Months and 6 Months
Population: Overall 13 pts consented for this study but 5 withdrew consent.
Measure: Mean (Standard Deviation); unit: mmHg/mm
Arm/Group | Baseline | Month 3 | Month 6
Number analyzed (Participants) | 8 | 8 | 8
mmHg/mm | 189.52 (41.19) | 225.82 (66.99) | 226.44 (44.07)

11. Secondary Outcome: Biomechanical Tissue Measurements (Energy Absorption)
Description: as for outcome 8
Time Frame: Baseline, 3 Months and 6 Months
Population: Overall 13 pts consented for this study but 5 withdrew consent.
Measure: Mean (Standard Deviation); unit: mmHg*mm
Arm/Group | Baseline | Month 3 | Month 6
Number analyzed (Participants) | 8 | 8 | 8
mmHg*mm | 74.32 (17.30) | 59.69 (15.78) | 61.04 (14.22)

12. Secondary Outcome: Change in Gene Expression
Description: Gene expression assessments will be completed to analyze protein related to collagen, elastin, and the extracellular matrix production. Gene Expression studies cellular activity and Collagen 1, Collagen 3, Elastin, LOX, IL8 and MMP2 are all biomarkers. Gene expression was only compared between baseline and 6 months.
  Fold changes were compared to control from Ct values of RT-qPCR reactions.
  * Ct: threshold cycle
  * RT-qPCR: Quantitative reverse transcription polymerase chain reaction)
Time Frame: Baseline and 6 Months
Measure: Mean (Standard Error); unit: fold change
Arm/Group | Month 6
Number analyzed (Participants) | 4
fold change
  Collagen 1 | 1.16 (0.28)
  Collagen 3 | 0.62 (0.42)
  Elastin | 1.72 (0.63)
  LOX | 1.06 (0.71)
  IL8 | 0.24 (0.18)
  MMP2 | 2.78 (1.98)

13. Secondary Outcome: Change in Histology Assessments
Description: Histological assessments (microscopic study-tissue structure, elastin, collagen and hyaluronic acid expression) will be completed after taking biopsies ( from the cheek adjacent to the nasolabial fold within the designated area for treatment) of the skin area to correlate changes to the skin after treatments. Histology studies the structure of the tissue. Collagen 3, Collagen 1, Elastin, Macrophage are biomarkers. Histology was only compared between baseline and 6 months.
  Fold changes compared to control were calculated from fluorescence intensity of a confocal microscopy images.
Time Frame: Baseline and 6 Months
Measure: Mean (Standard Error); unit: fold change
Arm/Group | Month 6
Number analyzed (Participants) | 6
fold change
  Collagen 3 | 37.82 (7.19)
  Collagen 1 | 7.22 (1.63)
  Elastin | 32.28 (5.98)
  Macrophage | 7.49 (1.73)

ADVERSE EVENTS:
Time Frame: Data was collected in a 6 month period after first treatment was completed
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT05085730/Prot_SAP_001.pdf